CLINICAL TRIAL: NCT02438423
Title: A Phase I Study of the Safety, Reactogenicity, Acceptability and Immunogenicity of Inactivated Influenza Vaccine Delivered by Microneedle Patch or by Hypodermic Needle
Brief Title: Inactivated Influenza Vaccine Delivered by Microneedle Patch or by Hypodermic Needle
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mark Prausnitz (Other)
Collaborators: Emory University (Other)
Responsible Party: Sponsor-Investigator, Mark Prausnitz, Investigator, Georgia Institute of Technology
Organization: Georgia Institute of Technology (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2015 TIV-MNP
Record Dates: First submitted 2015-05-06; First posted 2015-05-08 (Estimated); Results first posted 2019-07-05 (Actual); Last update posted 2019-07-05 (Actual); Status verified 2019-04

CONDITIONS: Influenza
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- IIV delivered by MN patch by study staff (Experimental): Inactivated influenza vaccine (IIV) delivered by microneedle (MN) patch administered by study staff
  Interventions: Biological: Inactivated influenza vaccine
- IIV delivered IM by study staff (Active Comparator): Inactivated influenza vaccine (IIV) delivered by intramuscular (IM) injection administered by study staff
  Interventions: Biological: Inactivated influenza vaccine
- IIV delivered by MN patch by subject (Experimental): Inactivated influenza vaccine (IIV) delivered by microneedle (MN) patch self-administered by subject
  Interventions: Biological: Inactivated influenza vaccine
- Placebo MN patch by study staff (Placebo Comparator): Placebo delivered by microneedle patch administered by study staff
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: Inactivated influenza vaccine — Seasonal trivalent inactivated influenza vaccine FDA-approved for 2014-2015 influenza season
  Arms: IIV delivered IM by study staff; IIV delivered by MN patch by study staff; IIV delivered by MN patch by subject
Other: Placebo
  Arms: Placebo MN patch by study staff

SUMMARY:
Title: A Phase I Study of The Safety, Reactogenicity, Acceptability and Immunogenicity of Inactivated Influenza Vaccine Delivered either by Microneedle Patch or by Hypodermic Needle.

This is a single center, partially blinded, randomized phase I study in which healthy adult subjects (ages 18-49) will receive either inactivated influenza vaccine (IIV) (either by microneedle patch or hypodermic needle) or placebo (by microneedle patch). This study is designed to investigate the safety, reactogenicity, acceptability and immunogenicity of an inactivated influenza vaccine delivered by microneedle patch.

DETAILED DESCRIPTION:
Title: A Phase I Study of The Safety, Reactogenicity, Acceptability and Immunogenicity of Inactivated Influenza Vaccine Delivered either by Microneedle Patch or by Hypodermic Needle.

Population: healthy adults, 18-49 years inclusive

Number of Sites: One

Study Duration: 12 months

Subject Duration: 6 months

Objectives:

Primary:

To evaluate the safety and reactogenicity following receipt of inactivated influenza vaccine delivered by microneedle patch (either by staff or self-administered).

Secondary:

To evaluate the HAI titers following receipt of inactivated influenza vaccine delivered either by microneedle patch or by hypodermic needle (both vaccines administered by study staff).

To evaluate unsolicited adverse events following receipt of IIV delivered by microneedle patch (administered by study staff or self-administered).

To evaluate new-onset chronic illnesses (NOCI) following receipt of IIV delivered by microneedle patch (administered by study staff or self-administered).

Exploratory:

To evaluate microneutralizing antibody titers following receipt of inactivated influenza vaccine delivered either by microneedle patch or by hypodermic needle (both vaccines administered by study staff).

To evaluate HAI +/- microneutralization and ELISA titers following receipt of inactivated influenza vaccine delivered by microneedle patch (administered by study staff or self- administered) and compare to inactivated influenza vaccine delivered by hypodermic needle (administered by study staff).

To evaluate HAI +/- microneutralization and ELISA titers following receipt of inactivated influenza vaccine delivered by microneedle patch (administered by study staff) and compare to inactivated Influenza vaccine delivered by microneedle patch (self-administered).

To evaluate T follicular helper cells following receipt of inactivated influenza vaccine delivered by microneedle patch (administered by study staff or self-administered) and compare to inactivated influenza vaccine delivered by hypodermic needle (administered by study staff).

To evaluate innate immunity signatures by microarrays following receipt of inactivated influenza vaccine delivered by microneedle patch (administered by study staff or self-administered) and compare to inactivated influenza vaccine delivered by hypodermic needle (administered by study staff).

To evaluate B memory cells, CD4 and CD8 central memory and effector T cells, intracellular cytokine staining (ICS) for interferon-gamma and interleukin-4, cross reactive T cells following receipt of inactivated influenza vaccine delivered by microneedle patch (administered by study staff or self- administered) and compare to inactivated influenza vaccine delivered by hypodermic needle (administered by study staff).

To evaluate the acceptability of inactivated Influenza vaccine delivered by microneedle patch (administered by study staff or self-administered) and compare to inactivated influenza vaccine delivered by hypodermic needle (administered by study staff).

Schematic of Study Design:

This is a single center, partially blinded, randomized phase I study in which healthy adult subjects (ages 18-49) will receive either inactivated influenza vaccine (IIV) (either by microneedle patch or hypodermic needle) or placebo (by microneedle patch). This study is designed to investigate the safety, reactogenicity, acceptability and immunogenicity of an inactivated influenza vaccine delivered by microneedle patch.

A total of 100 subjects (25 subjects in each group) will be randomized to one of four groups as in the schematic of the study design below.

Group A: Inactivated influenza vaccine delivered by microneedle patch administered by study staff Group B: Inactivated influenza vaccine delivered by intramuscular injection administered by study staff Group C: Inactivated influenza vaccine delivered by microneedle patch administered by subject Group D: Placebo delivered by microneedle patch and administered by study staff

Each subject will have 6 clinic visits: D0, D2 (+1 day), D8 (+2 days), D28 (+/- 2 days), D56 (+/- 5 days), and D180( +/- 14 days).

Blood draws will be obtained at 6 clinic visits to evaluate for immunogenicity (D0, D2 (+1 day) D8 (+ 2 days) - D28 (+/- 2 days), D56 (+/- 5 days), and D180 (+/- 14 days)) and at four clinic visits for safety (D0, D2 (+1 day), D8 (+2 days), and D28 (+/- 2 days)).

Safety will be measured by the occurrence of solicited injection site and systemic reactogenicity on the day of study product administration through 7 days after, and serious adverse events (SAEs) and new-onset chronic medical conditions through 180 days after study product administration.

Immunogenicity testing will include performing hemagglutination inhibition (HAI) +/- microneutralizing antibody assays as well as other adaptive immune assays on D0 prior to study product administration and at D8 (+2 days) , D28 (+/- 2 days), D56 (+/-5 days), and D180 (+/-14 days)) .

ELIGIBILITY:
Inclusion Criteria:

1. Subject provides written informed consent prior to any study procedures being performed.
2. Subject is male or non-pregnant female between the ages of 18 and 49, inclusive, on the day of signing informed consent.
3. Subject is in good health as determined by vital signs, medical history and targeted physical examination
4. Women of childbearing potential must agree to practice abstinence from sexual intercourse with men or use acceptable contraception, initiated at least 30 days prior to the study vaccination throughout D180 in order to avoid pregnancy.
5. Women of childbearing potential must have a negative urine pregnancy test prior to administration of the study product.
6. Subject is able to understand and comply with required study procedures.

Exclusion Criteria:

1. Subject has received a 2014-2015 seasonal influenza vaccine.
2. Subject with documented influenza infection during the 2014-2015 influenza season.
3. Subject has touched or handled a microneedle patch prior to study enrollment (excluding dermaroller-like devices).
4. Subject has a known allergy to eggs, egg or chicken protein or other components of the study product
5. Subject has a history of severe reactions following previous immunization with licensed influenza virus vaccines.
6. Subject has an acute illness with fever (temperature >100.4 °F) within 72 hours prior to vaccination.
7. Subject has a known chronic medical problem
8. Subject has known immunosuppression due to underlying illness or treatment
9. Subject has a scar, tattoo, rash or other dermatologic condition in the area of the vaccination site which will interfere with the assessment of injection site reactogenicity.
10. Subject has a history of keloid formation.
11. Subject has used long-term* high-dose** oral or parenteral glucocorticoids, or high-dose inhaled steroids***.

    * Long term is defined as taken for 2 weeks or more in total at any time during the past 2 months.
    * High dose defined as prednisone ≥ 20 mg total daily dose, or equivalent dose of other glucocorticoids.
    * High dose defined as > 800 mcg/day of beclomethasone dipropionate or equivalent.

    If short term corticosteroids are given, then the subject should not receive study vaccination or have blood collected for immunogenicity studies within 1 week of steroid administration
12. Subject has a history of Guillain-Barre Syndrome.
13. Subject is pregnant, post-partum (<12 months after delivery), or breast feeding or plans to breastfeed during the study.
14. Alcohol or drug abuse and psychiatric conditions that, in the opinion of the investigator, would preclude compliance with the trial or interpretation of safety or endpoint data.
15. Subject has any condition that, in the opinion of the investigator, may put the subject at increased risk of harm, may cause the subject to be unable to meet the requirements or might otherwise interfere with evaluations required by the study.
16. Subject has received any experimental products within 30 days before study entry or plan to receive experimental products at any time during the study.
17. Subject has received a live vaccine within 28 days prior to study entry or plans to receive a live vaccine prior to Day 28 of the study.
18. Subject has received an inactivated vaccine within 14 days prior to study entry or plans to receive an inactivated vaccine prior to Day 28 of the study.
19. Subject has received immunoglobulin or blood products in the past 90 days or planned receipt at any time during the study.
20. Subject BMI >35 kg/m2.
21. Subject has a systolic blood pressure >160 or < 80 mmHg or diastolic blood pressure >100 or < 60 mmHg.
22. Subject has a resting pulse rate < 50 bpm or >100 bpm.
23. Subject donated blood 56 days before screening OR will donate blood on or before day 28 of the study.

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2015-06; Primary Completion 2016-03-23 (Actual); Study Completion 2016-03-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nadine Rouphael, MD, Principal Investigator — Emory University
Locations (1):
- The Hope Clinic, Decatur, Georgia, United States

REFERENCES:
- [Derived] Rouphael NG, Paine M, Mosley R, Henry S, McAllister DV, Kalluri H, Pewin W, Frew PM, Yu T, Thornburg NJ, Kabbani S, Lai L, Vassilieva EV, Skountzou I, Compans RW, Mulligan MJ, Prausnitz MR; TIV-MNP 2015 Study Group. The safety, immunogenicity, and acceptability of inactivated influenza vaccine delivered by microneedle patch (TIV-MNP 2015): a randomised, partly blinded, placebo-controlled, phase 1 trial. Lancet. 2017 Aug 12;390(10095):649-658. doi: 10.1016/S0140-6736(17)30575-5. Epub 2017 Jun 27. PMID 28666680

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo MN Patch by Study Staff: Placebo delivered by microneedle patch administered by study staff
  Placebo
Period: Overall Study
Arm/Group | IIV Delivered by MN Patch by Study Staff | IIV Delivered IM by Study Staff | IIV Delivered by MN Patch by Subject | Placebo MN Patch by Study Staff
Started | 25 | 25 | 25 | 25
Completed | 25 | 25 | 25 | 25
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | IIV Delivered by MN Patch by Study Staff | IIV Delivered IM by Study Staff | IIV Delivered by MN Patch by Subject | Placebo MN Patch by Study Staff | Total
Number analyzed (Participants) | 25 | 25 | 25 | 25 | 100
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 25 | 25 | 25 | 25 | 100
  >=65 years | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 11 | 12 | 12 | 47
  Male | 13 | 14 | 13 | 13 | 53
Race/Ethnicity, Customized [Number; unit: participants] — Population: The different rows describe subsets of the population and the numbers add up to the overall number (100 subjects)
  participants
    White | 11 | 12 | 14 | 12 | 49
    Black | 8 | 8 | 8 | 7 | 31
    Other | 6 | 5 | 3 | 6 | 20

OUTCOME MEASURES:

1. Primary Outcome: Occurrence of Solicited Injection Site and Systemic Reactogenicity on the Day of Study Product Administration Through 7 Days After Administration.
Description: Safety will be measured by the occurrence of solicited injection site and systemic reactogenicity on the day of study product administration through 7 days after, and serious adverse events (SAEs) and new-onset chronic medical conditions through 180 days after study product administration. Local and systemic reactions were graded using an Injection Site Reaction table listing local reactions (e.g., swelling, erythema, etc.) and grade levels from 0 to 4 for each local reaction, a General Adverse Reaction table listing systemic reactions (e.g., fatigue, myalgia, etc.) and grade levels from 0 to 4 for each systemic reaction, and a Clinical Adverse Event Grading Scale (grades 1-4) for safety labs. In all tables, the higher the grade, the worse the adverse event.
Time Frame: From Day 0 through Day 8
Measure: Number; unit: Reactions
Arm/Group | IIV Delivered by MN Patch by Study Staff | IIV Delivered IM by Study Staff | IIV Delivered by MN Patch by Subject | Placebo MN Patch by Study Staff
Number analyzed (Participants) | 25 | 25 | 25 | 25
Reactions
  Reactions D1-D7 (pruritus) | 20 | 4 | 21 | 4
  Reactions D1-D7 (Pain) | 5 | 11 | 5 | 2
  Reactions D1-D7 (Redness/Erythema) | 10 | 0 | 10 | 0
  Reactions D1-D7 (Tenderness) | 17 | 15 | 16 | 4
  Reactions D1-D7 (Nausea) | 2 | 4 | 2 | 1
  Reactions D1-D7 (Fatigue) | 13 | 10 | 4 | 5
  Reactions D1-D7 (Headache) | 5 | 7 | 7 | 2
  Reactions D1-D7 (Swelling/Induration) | 4 | 1 | 2 | 0
  Reactions D1-D7 (Myalgia) | 4 | 7 | 1 | 4
  Reactions D1-D7 (Shivering/Shaking) | 1 | 2 | 0 | 1
  Reactions D1-D7 (Arthralgia) | 0 | 2 | 3 | 1
  Reactions D1-D7 (Fever) | 1 | 0 | 0 | 0
  Reactions D1-D7 (Malaise) | 4 | 5 | 0 | 1
  Reactions D1-D7 (Sweating) | 3 | 5 | 2 | 0

2. Primary Outcome: Occurrence of Study Product-related Serious Adverse Events From D0 Until D180 (+/- 14 Days) After Study Product Administration.
Time Frame: From Day 0 until Day 180
Measure: Number; unit: Serious adverse events
Arm/Group | IIV Delivered by MN Patch by Study Staff | IIV Delivered IM by Study Staff | IIV Delivered by MN Patch by Subject | Placebo MN Patch by Study Staff
Number analyzed (Participants) | 25 | 25 | 25 | 25
Serious adverse events | 0 | 0 | 0 | 0

3. Primary Outcome: Occurrence of Grade 3 Solicited or Unsolicited Adverse Events From D0 Until D28 (+/- 2 Days) After Study Product Administration.
Time Frame: From Day 0 until Day 28
Measure: Number; unit: Grade 3 adverse events
Arm/Group | IIV Delivered by MN Patch by Study Staff | IIV Delivered IM by Study Staff | IIV Delivered by MN Patch by Subject | Placebo MN Patch by Study Staff
Number analyzed (Participants) | 25 | 25 | 25 | 25
Grade 3 adverse events | 0 | 0 | 0 | 0

4. Secondary Outcome: Geometric Mean Titer (GMT) of HAI Antibody Approximately 28 Days Following Receipt of IIV Delivered by Microneedle Patch or by Hypodermic Needle (Both Vaccines Administered by Study Staff).
Time Frame: At Day 28
Measure: Geometric Mean (95% Confidence Interval); unit: HAI Antibody Titers (GMT)
Arm/Group | IIV Delivered by MN Patch by Study Staff | IIV Delivered IM by Study Staff
Number analyzed (Participants) | 25 | 25
HAI Antibody Titers (GMT)
  A/Christchurch (H1N1) | 1197 [854.6 to 1675] | 997.3 [703 to 1415]
  A/Texas (H3N2) | 287 [191.5 to 430.2] | 223.2 [159.8 to 311.7]
  B/Massachusetts | 125.8 [85.92 to 184.1] | 94.48 [73.5 to 121.5]

5. Secondary Outcome: Percentage of Subjects Achieving Seroprotection (Defined as a HAI Antibody Titer of 1:40 or Greater) Approximately 28 Days Following Receipt of IIV Delivered by Microneedle Patch or by Hypodermic Needle (Both Vaccines Administered by Study Staff).
Time Frame: At Day 28
Measure: Number (95% Confidence Interval); unit: percentage of subjects (seroprotected)
Arm/Group | IIV Delivered by MN Patch by Study Staff | IIV Delivered IM by Study Staff
Number analyzed (Participants) | 25 | 25
percentage of subjects (seroprotected)
  A/Christchurch (H1N1) | 100 [85.8 to 100] | 100 [86.3 to 100]
  A/Texas (H3N2) | 100 [85.8 to 100] | 100 [86.3 to 100]
  B/Massachusetts | 96 [78.9 to 99.9] | 100 [86.3 to 100]

6. Secondary Outcome: Percentage of Subjects Achieving Seroconversion Approximately 28 Days Following Receipt of IIV Delivered by Microneedle Patch or by Hypodermic Needle (Both Vaccines Administered by Study Staff).
Description: Seroconversion is defined as either a pre-vaccination HAI titer <1:10 and a post-vaccination HAI titer ≥1:40, or a pre-vaccination HAI titer ≥1:10 and a minimum four-fold rise in post-vaccination HAI antibody titer.
Time Frame: At Day 28
Measure: Number (95% Confidence Interval); unit: percentage of subjects who seroconverted
Arm/Group | IIV Delivered by MN Patch by Study Staff | IIV Delivered IM by Study Staff
Number analyzed (Participants) | 25 | 25
percentage of subjects who seroconverted
  A/Christchurch (H1N1) | 92 [73 to 99] | 80 [59.3 to 93.2]
  A/Texas (H3N2) | 83 [62.6 to 95.3] | 76 [54.9 to 90.6]
  B/Massachusetts | 71 [48.9 to 87.4] | 32 [15 to 53.5]

ADVERSE EVENTS:
Arm/Group | IIV Delivered by MN Patch by Study Staff | IIV Delivered IM by Study Staff | IIV Delivered by MN Patch by Subject | Placebo MN Patch by Study Staff
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/25 | 0/25 | 0/25
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/25 | 1/25 | 0/25
Other Adverse Events (participants affected / at risk) | 23/25 | 20/25 | 23/25 | 12/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IIV Delivered by MN Patch by Study Staff (N=25) | IIV Delivered IM by Study Staff (N=25) | IIV Delivered by MN Patch by Subject (N=25) | Placebo MN Patch by Study Staff (N=25)
Severe acute enteritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — severe acute enteritis (i.e. abdominal pain, nausea, and vomiting)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | IIV Delivered by MN Patch by Study Staff (N=25) | IIV Delivered IM by Study Staff (N=25) | IIV Delivered by MN Patch by Subject (N=25) | Placebo MN Patch by Study Staff (N=25)
Swelling/Induration (grade 1) (General disorders) | 4 | 1 | 1 | 0
Redness/Erythema (grade 1) (General disorders) | 9 | 0 | 8 | 0
Tenderness (grade 1) (General disorders) | 13 | 9 | 14 | 3
Pain (grade 1) (General disorders) | 5 | 8 | 4 | 2
Pruritis (itching) (grade 1) (General disorders) | 16 | 3 | 20 | 4
Fatigue (General disorders) | 12 | 7 | 2 | 5
Body ache (myalgia) (grade 1) (General disorders) | 4 | 6 | 1 | 3
Shivering/shaking body movements (grade 1) (General disorders) | 1 | 1 | 0 | 1
Sweating (grade 1) (General disorders) | 3 | 5 | 2 | 0
Malaise (grade 1) (General disorders) | 4 | 2 | 0 | 1
Nausea (grade 1) (General disorders) | 2 | 3 | 1 | 6
Fever (grade 1) (General disorders) | 1 | 0 | 6 | 0
Joint pain (arthralgia) (grade 1) (General disorders) | 0 | 1 | 2 | 1
Anemia (grade 1) (Blood and lymphatic system disorders) | 5 | 2 | 1 | 3
Decreased absolute lymphocytes (grade 1) (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Leukocytosis (grade 1) (Blood and lymphatic system disorders) | 1 | 1 | 0 | 0
Leukopenia (grade 1) (Blood and lymphatic system disorders) | 3 | 1 | 1 | 3
Thrombocytopenia (grade 1) (Blood and lymphatic system disorders) | 0 | 1 | 0 | 1
Gastroenteritis (grade 1) (Gastrointestinal disorders) | 2 | 0 | 0 | 0
Epigastric pain (grade 1) (Gastrointestinal disorders) | 0 | 0 | 0 | 1
URI (grade 1) (Infections and infestations) | 1 | 2 | 1 | 1
Elevated ALT (grade 1) (Investigations) | 1 | 0 | 0 | 2
Transaminitis (grade 1) (Investigations) | 0 | 0 | 0 | 1
Elevated CK (grade 1) (Investigations) | 0 | 1 | 0 | 0
Left elbow tendonitis (grade 1) (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Neck pain (grade 1) (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Arthralgia (grade 1) (Musculoskeletal and connective tissue disorders) | 0 | 1 | 2 | 1
Leg pain (grade 1) (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Headache (grade 1) (Nervous system disorders) | 0 | 6 | 6 | 0
Tooth infection (grade 1) (Infections and infestations) | 0 | 0 | 1 | 0
Toe infection (grade 1) (Infections and infestations) | 0 | 0 | 1 | 0
Conjunctivitis (grade 1) (Infections and infestations) | 0 | 0 | 1 | 0
Presyncope (grade 1) (Nervous system disorders) | 0 | 0 | 1 | 0
Hypertension (grade 1) (Vascular disorders) | 0 | 0 | 1 | 0
Elevated ALT AST (grade 1) (Investigations) | 0 | 0 | 1 | 1
Redness/Erythema (grade 2) (General disorders) | 1 | 0 | 2 | 0
Tenderness (grade 2) (General disorders) | 4 | 6 | 1 | 1
Pruritis (grade 2) (General disorders) | 3 | 1 | 1 | 0
Fatigue (grade 2) (General disorders) | 12 | 2 | 2 | 0
Pain (grade 2) (General disorders) | 0 | 3 | 1 | 0
Body ache (myalgia) (grade 2) (General disorders) | 0 | 1 | 0 | 1
Shivering/shaking Body Movements (grade 2) (General disorders) | 0 | 1 | 0 | 0
Malaise (grade 2) (General disorders) | 0 | 3 | 3 | 0
Joint pain (Arthralgia) (grade 2) (General disorders) | 0 | 1 | 1 | 0
Nausea (grade 2) (General disorders) | 0 | 1 | 1 | 1
Swelling/Induration (grade 2) (General disorders) | 0 | 0 | 1 | 0
Neutropenia (grade 2) (Blood and lymphatic system disorders) | 1 | 0 | 1 | 2
Thrombocytopenia (grade 2) (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Headache (grade 2) (Nervous system disorders) | 1 | 1 | 0 | 1
Vomiting (grade 2) (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Arthralgia (grade 2) (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Left hand bruise (grade 2) (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Hypertension (grade 2) (Vascular disorders) | 0 | 0 | 1 | 0
Pruritis (grade 3) (General disorders) | 1 | 0 | 0 | 0
Fatigue (grade 3) (General disorders) | 0 | 1 | 0 | 0
Elevated ALT (grade 3) (Investigations) | 0 | 1 | 0 | 0
Tenderness (grade 3) (General disorders) | 0 | 0 | 1 | 0
Acute enteritis (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Headache (grade 3) (Nervous system disorders) | 0 | 0 | 0 | 1
Hypertension (grade 3) (Vascular disorders) | 0 | 0 | 0 | 1
Elevated AST (grade 4) (Investigations) | 0 | 0 | 1 | 0
Elevated CK (grade 4) (Investigations) | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No